CLINICAL TRIAL: NCT02710292
Title: Clinical Evaluation of DAILIES TOTAL 1® in Japanese Population - Comparison of Lens Centration Between DAILIES TOTAL 1® and 1-DAY ACUVUE® TruEye®
Brief Title: Clinical Evaluation of DAILIES TOTAL 1® Performance in a Japanese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLS104-P001
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-05

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- DT1, then TE (Other): Delefilcon A contact lenses worn first, followed by narafilcon A contact lenses. Each product will be worn bilaterally (in both eyes) for at least 7 days in a daily disposable modality.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses
- TE, then DT1 (Other): Narafilcon A contact lenses worn first, followed by delefilcon A contact lenses. Each product will be worn bilaterally (in both eyes) for at least 7 days in a daily disposable modality.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses
  Other Names: DAILIES TOTAL 1®; DT1
Device: Narafilcon A contact lenses
  Other Names: 1-DAY ACUVUE® TruEye®

SUMMARY:
The purpose of this study is to compare DAILIES TOTAL1® (DT1) to 1-DAY ACUVUE® TruEye® (TE) for Investigator-rated successful lens centration in Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form;
* Habitual current daily disposable soft contact lenses wearer;
* Symptoms of contact lens discomfort as defined by the Symptomatology (Eligibility) Questionnaire;
* Lenses within the power range specified in the protocol;
* Vision correctable to 20/25 or 0.1 logMAR (logarithmic minimum angle of resolution) or better in each eye at distance with pre-study contact lenses at Visit1;
* Acceptable lens fit with both study contact lenses;
* Willing to wear lenses every day or at least for a minimum of 10 days, 6 hours per day, every day if possible and attend all study visits;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Currently wearing DT1 or TE sphere lenses;
* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications in which contact lens wear could be contraindicated as determined by the investigator;
* Eye injury or surgery within 12 weeks immediately prior to enrollment;
* History of herpetic keratitis, ocular surgery or irregular cornea;
* Prior refractive surgery;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Participation in any clinical trial within 30 days of the enrollment visit;
* Other protocol-specified exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Clinical Development, Study Director — Alcon Japan, Ltd.
Locations (1):
- Contact Alcon Japan, Ltd. for Trial Locations, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 study sites located in Japan.
Pre-assignment Details: Of the 104 subjects, 5 were exited as screen failures prior to being enrolled. This reporting group includes all enrolled subjects (99).
Period: Period 1, First 10 Days of Wear
Arm/Group | DT1, Then TE | TE, Then DT1
Started | 47 | 52
Completed | 46 | 49
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Period: Period 2, Second 10 Days of Wear
Arm/Group | DT1, Then TE | TE, Then DT1
Started | 46 | 49
Completed | 46 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who used the study device (Safety Analysis Set).
Groups:
- Overall: Delefilcon A and narafilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Investigator-rated Lens Centration of "Optimal" After 10 Days of Wear
Description: Lens centration was assessed by the investigator on a 5-point scale, where 0=Optimal and 4=Severe decentration (with corneal exposure). Both eyes contributed to the analysis.
Time Frame: Day 10, each product
Population: This analysis population includes all subjects who used the study device and in whom data after the use of the study device were available (Full Analysis Set).
Measure: Number; unit: percentage of subjects
Groups:
- Dailies Total1: Delefilcon A contact lenses worn bilaterally during Period 1 or Period 2 for for at least 7 days in a daily disposable modality.
- TruEye: Narafilcon A contact lenses worn bilaterally during Period 1 or Period 2 for at least 7 days in a daily disposable modality.
Arm/Group | Dailies Total1 | TruEye
Number analyzed (Participants) | 95 | 97
percentage of subjects | 89.5 | 47.4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 26 days). AEs are reported as pretreatment and treatment-emergent.
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device (test article). AE's were obtained as volunteered and elicited comments from the subjects and as observations by the Investigator.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- Dailies Total1: All subjects exposed to delefilcon A contact lenses
- TruEye: All subjects exposed to narafilcon A contact lenses
Arm/Group | Pretreatment | Dailies Total1 | TruEye
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/96 | 0/98
Other Adverse Events (participants affected / at risk) | 0/104 | 7/96 | 23/98
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=104) | Dailies Total1 (N=96) | TruEye (N=98)
Dry Eye (Eye disorders) | 0 | 5 | 5
Punctate keratitis (Eye disorders) | 0 | 2 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.